CLINICAL TRIAL: NCT00709644
Title: A Pivotal Bioequivalence Study of 250 Mcg NGM/25 Mcg EE With or Without Folic Acid in Healthy Female Subjects
Brief Title: Bioequivalence Study of the Oral Contraceptive (OC) Tablet Containing Norgestimate (NGM)/Ethinyl Estradiol (EE) With or Without Folic Acid in Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CR002203
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Pharmacokinetics; Therapeutic Equivalency; Contraceptives, Oral
Keywords: Ortho Tri-Cyclen Lo; Contraceptives, Oral; Norgestimate; Ethinyl Estradiol; Folic Acid; Female Contraception
MeSH Terms: interventions — norgestimate; Ethinyl Estradiol; Folic Acid

INTERVENTIONS:
Drug: Norgestimate; Ethinyl Estradiol; Folic acid.

SUMMARY:
The purpose of the study is to determine the bioequivalence of Norgestimate (NGM) and Ethinyl Estradiol (EE) in 2 formulations of 250 mcg NGM/25 mcg EE, 1 without folic acid and 1 containing 400 mcg folic acid. The pharmacokinetics of blood folate from the formulation of 250 mcg NGM/25 mcg EE containing 400 mcg folic acid and from 400 mcg folic acid administered alone is characterized.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized (study drug assigned by chance), 3-way crossover bioequivalence study of a single dose of 250 mcg NGM/25 mcg EE with or without folic acid. The study consisted of a pretreatment phase (a screening period lasting up to 21 days), an open-label treatment phase (consisting of 3 periods during which a single dose of study drug was administered followed by up to 72 hours of serial blood sample collections for pharmacokinetic analysis), and a posttreatment phase (consisting of safety evaluations at the completion of the third open-label treatment period or at early withdrawal). All healthy volunteers received the following treatments (1 during each period): Treatment A: 250 mcg NGM/25 mcg EE; Treatment B: 250 mcg NGM/25 mcg EE plus folic acid 400 mcg (combined formulation); Treatment C: folic acid 400 mcg. Healthy volunteers were randomly assigned to 1 of 6 treatment sequence groups (ABC, ACB, BAC, BCA, CAB, or CBA) on Day 1 of the first open-label treatment period. Healthy volunteers received a single dose of study drug on Day 1 in each period according to their assigned treatment sequence. There was a washout period between treatments of at least 4 weeks. Healthy volunteers were confined to the study unit from the evening before dosing (Day -1) until after vital signs were measured following collection of the 24-hour (Treatment C) or 48-hour (Treatments A or B) postdose blood sample. Blood samples were collected at specified times for 24 hours after dosing for the determination of plasma levels of folate and for 72 hours after dosing for the determination of blood levels of norelgestromin (NGMN), and norgestrel (NG) [the active breakdown products of NGM], and EE. Safety was evaluated based on the following: the incidence, type, and severity of adverse events; clinical laboratory tests; vital sign and electrocardiogram (ECG) measurements; and physical and gynecological (including breast) examinations. Oral temperature, heart rate, respiratory rate, and blood pressure were measured at screening, before each dose, and at least 15 minutes after the 24-hour (all treatments) and 48- and 72-hour (healthy volunteers who received Treatments A or B) pharmacokinetic blood samples in each period, or at early withdrawal. In Period 3, the end-of-study assessments were considered the 24-hour (for healthy volunteers who received Treatment C) and the 72-hour (for healthy volunteers who received Treatments A and B) measurements. Physical and gynecologic examinations and ECG were performed at screening, and at least 1 hour after the last pharmacokinetic blood sample on Day 58 for healthy volunteers who received Treatment C in Period 3, on Day 60 for healthy volunteers who received Treatments A or B in Period 3, or at early withdrawal. Blood samples for blood chemistry, hematology, and urine samples for urinalysis were collected at screening, after the last pharmacokinetic blood sample on Day 58 for healthy volunteers who received Treatment C in the third treatment period, on Day 60 for healthy volunteers who received Treatments A or B in Period 3, or at early withdrawal. The total duration of the study, not including the pretreatment phase, was approximately 9 weeks. Treatment A (250 mcg NGM/25 mcg EE) was administered as a single tablet corresponding to Days 15 to 21 in the commercial dialpak of the OC study drug; Treatment B (250 mcg NGM/25 mcg EE plus 400 mcg of folic acid) was administered as a single tablet; and Treatment C (400 mcg of folic acid) was administered as single United States Pharmacopoeia (USP) tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* nonpregnant
* nonlactating
* nonsmoking women
* weighing at least 110 pounds
* With regular menstrual cycles
* A body mass index between 16 and 29.9 kg/m2
* And a hematocrit of at least 36%.

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to sex hormonal therapy including: thromboembolic disorders cerebral vascular or coronary artery disease, chronic untreated hypertension, or migraines, benign or malignant liver tumor that developed during the use of OC
* Known or suspected estrogen-dependent neoplasia
* Presence of disorders commonly accepted as contraindications to combined OC including: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, or liver disease
* Intake any multivitamin or folic acid-containing supplements within 21 days before study admission
* Used a steroid hormone-containing intrauterine device within 3 months before study admission
* Used any medications that were known cytochrome P-450 enzyme inducers or inhibitors (e.g., St. John's Wort, cimetidine or rifampin), within 60 days before dosing.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2005-04; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Determine the bioequivalence of NGM (as measured by the pharmacokinetics of its active breakdown product NGMN) and EE in 2 formulations of 250 mcg NGM/25 mcg EE, 1 without folic acid and 1 containing 400 mcg folic acid.

SECONDARY OUTCOMES:
Determine the pharmacokinetics of NG in these 2 formulations; and to characterize the pharmacokinetics of plasma folate after the administration of folic acid alone or in combination with 250 mcg NGM/25 mcg EE. Safety also was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Bioequivalence study of the oral contraceptive tablet containing norgestimate (250 mcg)/ethinyl estradiol (25 mcg) with or without folic acid in healthy women. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=455&filename=CR002203_CSR.pdf